CLINICAL TRIAL: NCT04123613
Title: A Multi-Center Open-label Investigation to Assess the Safety and Efficacy of Multiple Doses of DM199 in Patients With Chronic Kidney Disease
Brief Title: Multiple Doses of DM199 in Patients With Chronic Kidney Disease (REDUX)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: DiaMedica Therapeutics Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DM199-2019-001
Record Dates: First submitted 2019-10-08; First posted 2019-10-11 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Kidney Diseases
MeSH Terms: conditions — Kidney Diseases | interventions — DM199

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 2.0 µg/kg, multiple dose (Experimental): n=45 with 15 Participants from cohort 1, 15 from cohort 2, and 15 from cohort 3
  Interventions: Drug: DM199
- 5.0 µg/kg, multiple dose (Experimental): n=45 with 15 Participants from cohort 1, 15 from cohort 2 and 15 from cohort 3
  Interventions: Drug: DM199

INTERVENTIONS:
Drug: DM199 — A pharmaceutical formulation comprised of recombinant human tissue kallikrein-1 (rhKLK-1) that is being developed as an injectable protein drug

SUMMARY:
An open-label, Phase II, multi-center study evaluating multiple doses of DM199 in participants with chronic kidney disease.

DETAILED DESCRIPTION:
This is an open-label, Phase II, multi-center study evaluating DM199 in approximately 90 Participants in three cohorts.

Cohort I: African Americans with CKD (Stage II or III), hypertension and non-diabetic Cohort II: Participants with IgA nephropathy diagnosis and CKD (Stage II or III) Cohort III: Diabetes Mellitus (Type II) with CKD (Stage II or III) and hypertension

Participants in each cohort will be enrolled in a parallel assignment to one of two doses:

Dose 1: DM199 2.0 µg/kg SC 2x week for 95 days Dose 2: DM199 5.0 µg/kg SC 2x week for 95 days

ELIGIBILITY:
Inclusion Criteria:

Cohort I

* African American
* Hypertension as defined by the American Heart Association for Stage I hypertension where systolic blood pressure (BP) ≥130 mmHg or diastolic BP ≥ 80 mmHg or on medication for treatment of hypertension.

Cohort II

* IgA nephropathy confirmed by medical history with biopsy

Cohort III

* Diabetes Mellitus (Type 2) with hypertension where systolic blood pressure (BP) ≥130 mmHg or diastolic BP ≥ 80 mmHg or on medication for treatment of hypertension
* Hemoglobin A1c ≥7% at screening

Both Cohorts

* Participant is willing and able to provide informed consent for study participation
* Participant male or female ≥ 18 years of age
* Participant has CKD as defined by using CKD EPI for Stage II 60 to <90 mL/min/1.73 m2 or Stage III 30 to <60 mL/min/1.73 m2
* UACR >150 mg/g and <5000 mg/g at screening
* Participant is clinically stable with respect to underlying renal impairment as assessed by the Investigator's medical evaluation

Exclusion Criteria:

* Participant has positive drug test for drugs of abuse and/or positive alcohol breath test at screening and Day 1
* Participant has a current diagnosis and/or is taking medication or diet control for diabetes (cohort I and II only)
* Participant has an A1c > 7% at screening (cohort I and II only)
* Participant received corticosteroid therapy within last 3 months
* Participant is unable or unwilling to comply with protocol requirements, including assessments, tests, and follow-up visits
* Participant has a history of significant allergic diathesis such as urticaria, angioedema, or anaphylaxis
* Participant has been previously diagnosed with kidney disease other than for hypertension, IgA or Diabetes Mellitus (Type II)
* Participant has hypotension as defined by systolic blood pressure ≤ 90 mmHg and diastolic blood pressure ≤ 60 mmHg at screen
* ACEi or GLP-1 medication prescribed for and taken by Participant (must not be taking for 5 half-lives prior to study drug administration and for 10 days post study drug administration)
* Participant has a current malignancy or active malignancy ≤ 2 years prior to enrollment except basal cell or squamous cell carcinoma of the skin or in situ cervical cancer that has undergone potentially curative therapy and ≥ 6 months have elapsed since the procedure
* Participant has an active infection at the time of enrollment, and/or a history of clinically significant acute bacterial, viral, or fungal systemic infections that required systemic treatment with a completed therapy in the last 7 days prior to enrollment
* Participant has known medical history of alpha 1-antitrypsin deficiency (α1-antitrypsin deficiency)
* Participant is pregnant or nursing or is planning a pregnancy during the study period
* Participant is male or female of childbearing potential, is participating in sexual activity that could lead to pregnancy and is unable or unwilling to practice medically effective contraception during the study
* Participant has received any investigational drug or device within 14 days (or 5 half lives, whichever is longer) prior to study drug administration starting on Day 1
* Participant has renal artery stenosis as determined at screen with medical history
* Participant received a kidney transplant
* Participant does not have adequate venous access for blood sampling
* Participant has any other medical condition which, in the opinion of the Investigator, will make participation medically unsafe or interfere with the study results
* Participant has any other clinically significant abnormalities in laboratory test results at screening that would, in the opinion of the Investigator, increase the Participant's risk of participation, jeopardize complete participation in the study, or compromise interpretation of study data
* Participant has any significant arrhythmia or conduction abnormality, which in the opinion of the Investigators and Medical Monitor may interfere with the safety of the Participant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2019-12-17 (Actual); Primary Completion 2022-03-16 (Actual); Study Completion 2022-03-16 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment emergent adverse events | 12 weeks
  Incidence, severity, and causality of adverse events
Change in renal function | 12 weeks
  eGFR
Change in urine albumin to creatinine ratio | 12 weeks
  UACR change from baseline
Plasma measurements of DM199 | 12 weeks
  Maximum plasma concentration of DM199

SECONDARY OUTCOMES:
Tumor necrosis factor receptor 1 (TNF R1) concentration in plasma, change from baseline | 12 weeks
  TNF R1 change from baseline
C-reactive protein (CRP) concentration in plasma, change from baseline | 12 weeks
  CRP change from baseline
Matrix metalloproteainase-9 (MMP-9) concentration in plasma, change from baseline | 12 weeks
  MMP-9 change from baseline
Vascular endothelial growth factor (VEGF) concentration in plasma, change from baseline | 12 weeks
  VEGF change from baseline
Cystatin C concentration in plasma, change from baseline | 12 weeks
  Cystatin C change from baseline
Prostaglandin E2 concentration in plasma, change from baseline | 12 weeks
  Prostaglandin E2 change from baseline
Prostacyclin concentration in plasma, change from baseline | 12 weeks
  Prostacyclin change from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Harry Alcorn, Pharm.D., Study Director — DiaMedica Inc.
Locations (14):
- United States (14):
  - Aventiv Research, Mesa, Arizona
  - Amcis Research Center, Granada Hills, California
  - IMD Clinical Trials Inc, Los Angeles, California
  - Amicis Reserch Center, Northridge, California
  - Innovative Healthcare Institute, Coral Springs, Florida
  - Elixia at Florida Kidney Physicians-SE, Fort Lauderdale, Florida
  - Pines Clinical Research-Hollywood, Hollywood, Florida
  - Elixia at Florida Kidney Physicians, Temple Terrace, Florida
  - Boise Kidney & Hypertension Institute, Meridian, Idaho
  - Research by Design LLC, Chicago, Illinois
  - New Orleans Center for Clinical Research, an AMR Company, New Orleans, Louisiana
  - Elixia At Clincal Renal Associates, Upland, Pennsylvania
  - Nephrotex Research Group, LLC, Dallas, Texas
  - RDRI, DeSoto, Texas

IPD SHARING:
Plan to Share IPD: No